CLINICAL TRIAL: NCT05989737
Title: A Randomized Controlled Trial of a AEBT Website for Adults With Skin Picking
Brief Title: A RCT of an AEBT Website for Adults With Skin Picking
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Utah State University (Other)
Responsible Party: Principal Investigator, Michael Twohig, Ph.D., Professor, Utah State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13693
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Excoriation (Skin-Picking) Disorder
Keywords: Acceptance and commitment therapy (ACT); Acceptance-enhanced behavioral training (AEBT)
MeSH Terms: conditions — Excoriation Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AEBT online program (Experimental): Participants will complete the 8-module intervention of Acceptance-enhanced behavior therapy (AEBT). Acceptance-enhanced behavior therapy is a manualized treatment approach created by Woods and Twohig 2008 that provides both Acceptance and Commitment Therapy and Habit Reversal Therapy.
  Interventions: Behavioral: Acceptance-Enhanced Behavior Therapy
- Waitlist control (No Intervention): Waitlist condition; only assessment

INTERVENTIONS:
Behavioral: Acceptance-Enhanced Behavior Therapy — 8-module intervention delivering acceptance-enhanced behavior therapy through a fully automated website. This intervention was adapted from the Acceptance-enhanced behavior therapy workbook (Woods & Twohig, 2008).
  Arms: AEBT online program

SUMMARY:
The goal of this clinical trial is to test an online intervention for adults with excoriation disorder (skin picking). The main questions it aims to answer are:

1. Is the online intervention effective, compared to a waitlist control condition?
2. Is the online intervention acceptable to use?

Participants will be randomized into either the online intervention or waitlist control condition:

1. Participants in the intervention condition will be asked to complete an 8 module acceptance-enhanced behavioral training (AEBT) program for skin picking and 4 surveys over 3 months.
2. Participants in the waitlist condition will be asked to complete 4 surveys over 3 months, and will receive access to the intervention once the study is complete.

DETAILED DESCRIPTION:
Excoriation disorder, also known as skin picking, is a chronic repetitive condition that impacts an individual's daily functioning and causes clinically significant distress. Excoriation is estimated to impact between 2-5% of the general population, although some studies have found up to 14% prevalence rates in undergraduate samples. Acceptance-enhanced behavioral training (AEBT), has shown promising results for targeting skin picking symptoms. However, a recent study demonstrated that mental health providers have limited knowledge of skin picking and how to treat it effectively, creating a dearth of available treatment opportunities .

This study aims to address the gap in accessible evidence-based excoriation treatment by examining the efficacy and feasibility of a self-guided, online program based in AEBT. Participants will be recruited from across the United States from August to November 2023, and will be randomized into either the online intervention group or a waitlist control condition. All participants will complete online self-report assessments at baseline, mid-, post-intervention, and 1 month follow-up, and waitlist participants will be provided access to the program once the study is complete. For the primary aim evaluating efficacy, the investigators predict that both primary (skin picking severity) and secondary outcomes (psychological flexibility, well-being, and distress) will be significantly improved in the active treatment condition compared to a waitlist control group. For the secondary aim evaluating feasibility, the investigators predict that participants will report acceptable feasibility as measured through treatment adherence, reports of usability, and program feedback.

ELIGIBILITY:
Inclusion Criteria:

* currently meet criteria for DSM-5 excoriation disorder
* at least 18 years old at intake
* fluent in English
* reside in the United States

Exclusion Criteria:

* currently receiving alternative psychotherapy for skin picking
* modifying or starting psychotropic medication 30 days prior to starting the study
* currently living outside of the United States
* under the age of 18
* did not meet DSM-5 criteria for excoriation at the time of intake session

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Skin Picking Scale - Revised (SPS-R) | 12 weeks
  The Skin Picking Scale - Revised is an 8-item self-report measure designed to assess skin picking severity over the past week. Items (e.g., "How often do you feel the urge to pick your skin?") are rated on a 5-point Likert Scale with total scores ranging from 0-32. Higher scores indicate greater skin picking severity.

SECONDARY OUTCOMES:
Acceptance and Action Questionnaire for Skin Picking (AAQ-SP) | 12 weeks
  The Acceptance and Action Questionnaire for Skin Picking is a 9-item (e.g., "I am able to not pick when the urge to pick is strong") self-report measure where items are rated from 1 (never true) to 7 (always true). Total scores range from 7-63 where lower scores indicate greater psychological flexibility around skin picking.
Depression Anxiety Stress Scale (DASS-21) | 12 weeks
  The Depression Anxiety Stress Scale is a 21-item self-report measure that assess general distress with three subscales: depression, anxiety, and stress. Items (e.g., "I found it difficult to relax") are rated from 0 (never) to 3 (almost always) on a 4-point Likert scale. Sum scores are calculated by adding the subscale items and multiplying by two, so total scores range from 0 to 120, with higher scores indicating more distress.
Mental Health Continuum-Short Form (MHC-SF) | 12 weeks
  The Mental Health Continuum Short Form is a 14-item self-report measure assessing emotional, social, and psychological well-being. Items (e.g., "During the past month, how often do you feel satisfied with life?") are rated from 0 (never) to 5 (everyday) on a 6-point Likert Scale. Total scores range from 0 to 70 where higher scores indicate greater levels of positive well-being.
The System Usability Scale (SUS) | 8 weeks
  The System Usability Scale measures the usability of technology-based systems using a 10-item self-report measure. Items are rated from 1 (strongly disagree) to 5 (strongly agree), and items will be modified to refer to self-help website for excoriation. Scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100; higher scores indicate better usability.
Treatment Evaluation Inventory-Short Form (TEI-SF) | 8 weeks
  The TEI-SF assesses treatment acceptability using a 9-item self-report measure. One item will be modified to refer to "skin picking" rather than "anxiety", as done in previous studies. Items are rated from 1 (strongly disagree) to 5 (strongly agree); total scores range from 9-45 with higher scores indicating more positive treatment evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Utah State University, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: No